CLINICAL TRIAL: NCT00802490
Title: Pilot Trial of a Brain-computer Interface System Based Programme for the Treatment of ADHD
Brief Title: Effectiveness of a Electroencephalogram (EEG) Biofeedback for the Treatment of ADHD
Acronym: EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Collaborators: Institute for Infocomm Research (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Lim Choon Guan, Consultant, National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSRB-A/07/472; NHG Grant: SIG 08/018; AV/SW/581/1107/I2R agreement
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Electroencephalogram biofeedback; Inattention; Brain-Computer Interface System
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): 20 sessions of EEG biofeedback training
  Interventions: Device: Brain-Computer Interface System
- Control (Placebo Comparator): Only 1 session of EEG biofeedback training
  Interventions: Device: Brain-Computer Interface System

INTERVENTIONS:
Device: Brain-Computer Interface System — Newly-developed video games employing neurofeedback strategy to be played twice a week, 1 hour per session for a period of ten weeks.
  Other Names: Neurobiofeedback; EEG biofeedback
  Arms: Intervention
Device: Brain-Computer Interface System — Newly-developed video games employing neurofeedback strategy to be played once for 1 hour.
  Arms: Control

SUMMARY:
The aim of this study is to investigate if electroencephalogram (EEG) biofeedback incorporating the use of video games is effective in improving inattentive symptoms in children with ADHD.

DETAILED DESCRIPTION:
This study will enroll 20 outpatient subjects aged 7 to 12 newly diagnosed with ADHD who have never received treatment with medication. These children should have inattentive symptoms, i.e. diagnosed with combined or inattentive subtype of ADHD, and should not have any of the exclusion criteria. Based on the gender ratios from other studies, we will enroll 8 boys and 2 girls into the intervention group, giving a male:female ratio of 4:1. 10 will be in the 'intervention' group and 10 in the 'control' group.

Informed consent will be obtained from the parents, and assent from the subjects, prior to any form of assessment or intervention as part of the study.

INTERVENTION

The 10 subjects in the intervention group will take part in a total of 20 sessions spread over a 10-week period. Each subject will first need to master a simple concentration task involving a fishing game. After this, the child will go on to play a second soccer game. Each game employs the BCI system, and is controlled by the child's concentration, which is fed to the computer via the EEG leads. The child watches the game on a computer screen. Each session may take approximately thirty minutes.

The other 10 children in the comparison group will act as controls. At the clinic visit at baseline assessment, they will play the fishing game. There will be no further intervention subsequently.

ASSESSMENT

The following questionnaires will be administered to all subjects in both study groups at week 5, week 10, and at 3 months post-intervention (week 22):

1. ADHD Rating Scale: parents and teachers
2. Child Behaviour Checklist (CBCL): parents
3. Teacher's Report Form (TRF): teachers

In addition, for those subjects in the intervention group, they will be given 2 worksheets (1 Maths and 1 short comprehension exercise) at the end of the intervention during visits 2, 4, 6, 8, 10, 12, 14, 16, 18 and 20 over the 10-week period. Their EEG activity will be recorded during the completion of these worksheets.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV-TR criteria for ADHD (Combined OR Inattentive subtype)

Exclusion Criteria:

* Present or history of medical treatment with stimulant medication and/or Atomoxetine
* Co-morbid severe psychiatric condition or known sensori-neural deficit, e.g. complete blindness or deafness
* History of epileptic seizures
* Known mental retardation (i.e. IQ 70 and below)
* Predominantly hyperactive/impulsive subtype of ADHD

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Reliable Change Index (RCI)on ADHD Rating Scale | week 0, 5, 10, 22

SECONDARY OUTCOMES:
CBCL Attention Problem Score Change | Week 5, 10, 22

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SS Fung, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health/Woodbridge Hospital, Singapore, Singapore, Singapore